CLINICAL TRIAL: NCT05776147
Title: Radiotherapy With Extreme Hypofractionation in Patients With Breast Cancer in Brazil: a Retrospective Cohort Study
Acronym: RADIANT
Status: Recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0122
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Radiotherapy Side Effect
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The radiotherapy scheme with extreme hypofractionation has gained space in clinical practice and, therefore, it is necessary to analyze the Brazilian national experience in selected patients with breast cancer, with the aim of evaluating the oncological outcomes and toxicities with the use of this treatment protocol.

DETAILED DESCRIPTION:
All patients diagnosed with breast cancer who meet the eligibility criteria at participating centers will be included. Data will be collected from medical records at selected centers. Data collection will start from the location activation date. Data from up to 500 patients are expected to be collected at centers across Brazil.

Patients recruited for this study will be identified at participating centers. Data on clinical, demographic and socioeconomic variables will be collected, as well as data on treatments performed and outcomes.

The patient data sources will be the patients' medical records. Patients will continue to receive treatment and clinical evaluations for their illness as determined by their medical team, in accordance with the standards of care and usual clinical practice at each center. No intervention is proposed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old;
* Diagnosis of breast cancer of any molecular subtype;
* Undergoing extreme hypofractionated radiotherapy (5 x 5.2Gy) postoperatively;
* Treated from December/2019 onward;
* With clinical and treatment data available in medical records.

Exclusion Criteria:

* The protocol does not provide exclusion criteria.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer undergoing radiotherapy with extreme hypofractionation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence | 18 months
  To evaluate the effectiveness of the extreme hypofractionation scheme, in 5 fractions of 5.2 Gy, in women with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Nader Marte, Principal Investigator — Latin American Cooperative Oncology Group
Locations (11):
- Brazil (11):
  - ICC - Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Hospital Sírio-Libanês DF, Brasília, Federal District
  - Hospital Márcio Cunha da Fundação São Francisco Xavier (HMC-FSFX), Ipatinga, Minas Gerais
  - Oncominas - Clínica de Oncologia no Sul de Minas, Pouso Alegre, Minas Gerais
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Instituto COI - Clínicas Oncológicas Integradas (Instituto Américas RJ), Rio de Janeiro
  - Hospital Sírio-Libanês SP, São Paulo
  - HAOC - Hospital Alemão Oswaldo Cruz, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - A.C. Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: No